CLINICAL TRIAL: NCT00006222
Title: A Phase I Trial of EMD 121974 in Patients With HIV Related Kaposi's Sarcoma
Brief Title: EMD 121974 in Treating Patients With HIV-Related Kaposi's Sarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02358; AMC-023; CDR0000068142 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-09-11; First posted 2004-05-26 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2001-04

CONDITIONS: Sarcoma
Keywords: AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi | interventions — Cilengitide

ARMS (1):
- Arm I (Experimental): Patients receive EMD 121974 IV twice a week for four weeks. Courses repeat every 4 weeks in the absence of disease progression. Cohorts of 3-6 patients receive escalating doses of EMD 121974 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose limiting toxicities.
  Interventions: Drug: cilengitide

INTERVENTIONS:
Drug: cilengitide

SUMMARY:
Phase I trial to study the effectiveness of EMD 121974 in treating patients who have HIV-related Kaposi's sarcoma. EMD 121974 may stop the growth of Kaposi's sarcoma by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety and toxicity of EMD 121974 in patients with HIV related Kaposi's sarcoma.

II. Determine the antiangiogenic activity of this drug in these patients. III. Determine the antitumor activity of this drug in these patients. IV. Determine the effect of this drug on CD4 and CD8 cell counts and percentages, and on HIV viral load in these patients.

V. Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is a dose escalation study.

Patients receive EMD 121974 IV twice a week for four weeks. Courses repeat every 4 weeks in the absence of disease progression. Cohorts of 3-6 patients receive escalating doses of EMD 121974 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose limiting toxicities.

Patients are followed for at least 1 month.

PROJECTED ACCRUAL: A total of 18-30 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven Kaposi's sarcoma
* Systemic chemotherapy not required
* Minimum of 2 lesions amenable to biopsy
* Measurable or evaluable disease HIV positive

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: Karnofsky 70-100%
* Life expectancy: At least 3 months
* Hemoglobin at least 8.0 g/dL
* Absolute neutrophil count at least 750/mm3
* Platelet count at least 75,000/mm3
* PT/PTT normal Bilirubin normal (bilirubin no greater than 3.5 mg/dL if secondary to indinavir therapy, provided direct bilirubin no greater than upper limit of normal (ULN))
* AST (SGOT) no greater than 2.5 times ULN
* Creatinine no greater than 1.5 mg/dL OR creatinine clearance at least 60 mL/min
* No prior ischemic coronary artery disease including prior myocardial infarction
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study
* No concurrent active infection (nonsystemic infection, e.g., herpes simplex, oral thrush, or warts, allowed)
* No gastric or duodenal ulcer within past 6 weeks unless healed

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior antineoplastic biologic therapy and recovered
* At least 3 weeks since prior myeloid growth factor
* Growth factors and transfusion allowed if dose requirement is stable for 4 weeks prior to therapy
* At least 2 weeks since prior chemotherapy (6 weeks since prior nitrosourea or mitomycin) and recovered
* Concurrent hydroxyurea as antiretroviral therapy allowed if dose stable for 4 weeks prior to study
* No concurrent systemic cytotoxic chemotherapy
* Recovered from prior endocrine therapy
* At least 2 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy
* At least 3 weeks since major surgery or 10 days since minor surgery and recovered
* At least 4 weeks since prior experimental therapy for Kaposi's sarcoma and recovered
* At least 2 weeks since prior local therapy to any indicator lesion
* No concurrent investigational drugs (except antiretroviral therapy)
* At least 2 weeks since prior acute treatment for infection or other serious medical illness
* Antiretroviral therapy must be stable for 4 weeks prior to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-09; Primary Completion 2001-03 (Actual); Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Klencke, MD, Study Chair — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Vanderbilt Cancer Center, Nashville, Tennessee